CLINICAL TRIAL: NCT06367556
Title: Emotion and Symptom-Focused Engagement (EASE) for Caregivers: A Phase III Randomized Controlled Trial of an Intervention Targeting Traumatic Stress in Parents of Children With Cancer
Brief Title: Emotion and Symptom-Focused Engagement (EASE) for Caregivers
Acronym: EASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Hospital for Sick Children (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Gary Rodin Research Team, Senior Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4542
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Trauma and Stressor Related Disorders; Pediatric Cancer; Caregiver Burden
MeSH Terms: conditions — Trauma and Stressor Related Disorders; Neoplasms; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Quantitative outcome assessors and data analysts will be blinded to participant treatment group. Blinding is not possible for trial participants, intervention providers, or pediatric oncology teams, as assignment cannot be hidden from these individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants randomized to the intervention group will receive the Emotion and Symptom-focused Engagement (EASE) intervention and usual care. EASE consists of 8-12 psychotherapeutic sessions (~30-60 minutes each) delivered by a trained mental health clinician over 12 weeks.
  Interventions: Behavioral: Emotion and Symptom-Focused Engagement (EASE)
- Usual Care (No Intervention): Participants randomized to the control group will receive usual care.

INTERVENTIONS:
Behavioral: Emotion and Symptom-Focused Engagement (EASE) — EASE sessions are directed to provide relational support, affect regulation, and problem-solving related to cancer in the child, to changes in spousal, family, and other relationships, and to the burden of multiple individual and family responsibilities.
  Arms: Treatment

SUMMARY:
The goal of this Phase III randomized controlled trial is to evaluate the effectiveness of a novel psychotherapeutic intervention called Emotion and Symptom-focused Engagement (EASE) in parents caring for a child or adolescent with cancer. The main question it aims to answer is:

- Is EASE plus usual care associated with less severe traumatic stress symptoms over six months, measured by area under the curve, when compared to usual care alone in the parents of children diagnosed with cancer in the preceding six months?

For the primary outcome analysis, area under the curve will be calculated for each participant. The statistical significance of the difference between arms will also be evaluated. Participants in both groups will complete questionnaires package at enrolment, and 4, 8, and 12 weeks, and 6 months after enrolment. They will also be invited to participate in optional qualitative interviews to better understand their experience.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified primary family caregiver/guardian (i.e., parent assuming the majority of care activities) of a child: i) <18yo; ii) diagnosed with a new or relapsed life-threatening cancer within the preceding six months (disease-type eligibility per the Pediatric Oncology Group of Ontario Networked Information System); and iii) receiving active cancer therapy;
* Age ≥18 years; and,
* Able to complete outcome measures and engage in EASE in English, which need not be their first language.

Exclusion Criteria:

* Impairment in cognitive functioning or communication that would preclude participation in EASE sessions or outcome measure completion, as determined by the research team;
* Receiving formal ongoing psychotherapy at the time of recruitment;
* Active suicidal intention, based on an item in the Distress Assessment and Response Tool (DART) that has been widely used in suicidal intention screening in cancer; or,
* Child not expected to survive past the duration of trial, as determined by the child's medical team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
The Stanford Acute Stress Reaction Questionnaire [SASRQ] | 6-months
  SASRQ is a 30-item self-report measure with a rating scale of 0-30 (total range 0-150) that assesses the presence and severity of traumatic stress symptoms. Higher scores reflect greater severity.

SECONDARY OUTCOMES:
The PTSD Checklist for DSM-5 [PCL-5] | 6-months
  PCL-5 is a 20-item self-report measure with a rating scale of 0-4 (total range 0-80) that assesses the presence and severity of traumatic stress symptoms. Higher scores reflect greater severity.
The SF-36v2 Health Survey | 6-months
  SF-36v2 consists of eight scales yielding two summary measures: physical and mental health. It can be scored using both norm-based scoring (NBS) algorithms and the original 0-100 scoring system, where higher scores indicate better health status.
Patient Health Questionnaire [PHQ-9] | 6-months
  PHQ-9 is a 9-item measure with a rating scale of 0-3 (total range 0-27) that assesses the presence and severity of depressive symptoms. Higher scores reflect greater depression severity.
Caregiver Self-Efficacy in Contributing to Patient Self Care Scale [CSE-CSC] | 6-months
  CSE-CSC is a 10-item scale (standardized score 0-100) of to measure the extent of self-efficacy of the caregiver when contributing to patient self-care in the complex care context. Higher scores indicate higher self-efficacy.
Family Adaptability and Cohesion Evaluation Scales III [FACES-III] | 6-months
  FACES-III is a 20-item measure with a rating scale of 1-5 that will be used to assess parent perceived family functioning. 10-items measure family cohesion and 10-items measure adaptability (range 10-50, respectively), with higher scores for each domain indicating greater connectivity or flexibility compared to disengagement or rigidity.
Clinical Evaluation Questionnaire [CEQ] | 6-months
  CEQ is a 7-item patient-reported experience measure with a rating scale of 0-4 that will assess the perceived benefits that caregivers experience in their interactions with healthcare providers in domains relevant to advanced cancer. A total score is calculated by summing the item scores where higher scores reflect greater perceived benefit.
Family Satisfaction with End-of-Life Care Tool, 10-item version [FAMCARE-10] | 6-months
  FAMCARE-10 was developed to measure family caregiver satisfaction with the care of patients with advanced cancer with a rating scale of 0 (dissatisfied) to 2 (satisfied) where higher total scores reflect greater satisfaction.

OTHER OUTCOMES:
Caregiver Reaction Assessment Scale [CRA] | 6-months
  CRA is a 24-item scale that measures the impact of providing care at the subscale level, with no overall summative score. Items have a rating scale of 1 (strongly disagree) to 5 (strongly agree) with five subscales that assess impact on schedule (/25), impact on finances (/15), lack of family support (/25), impact on health (/20), and self-esteem (/30).The items in four of the scales (all except self-esteem) are generally phrased in a negative connotation such that higher scores indicate a more negative experience for that subscale.
ENRICHD Social Support Instrument [ESSI] | 6-months
  ESSI is a 7-item scale used to measure perceived social support. The first six items have a rating scale of 1 (none of the time) to 5 (all of the time) and the seventh is scored 4 for 'yes' and 2 for 'no'. Total scores range from 8 to 34. A lower total score reflects less support.
Experiences in Close Relationships Scale [ECR-16] | 6-months
  ECR-16 will be used to measure attachment security with a rating scale of 1 (disagree) to 7 (agree) with two subscales: Attachment Anxiety and Attachment Avoidance. Both subscales have a total score of 56 where higher scores indicate high attachment insecurity.
Hope of Improvement subscale of the Therapy Expectation and Evaluation Scale [PATHEVH] | Baseline
  This 4-item subscale (items 1, 4, 5, and 9) will be used to assess expectation of the effectiveness of Emotion and Symptom-focused Engagement (EASE) in the treatment arm. They are rated from 1 (absolutely wrong) to 5 (absolutely right) and items 1, 5, and 9 are reversed-scored prior to summing all items (total score range 4-20) with higher scores reflecting more positive outcome expectation.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Princess Margaret Cancer Centre - University Health Network, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No